CLINICAL TRIAL: NCT07220928
Title: The Effect of a Cold Air Eucapnic Hyperventilation Test on Lower Respiratory Airways in Healthy Volunteers and Patients With Asthma
Acronym: CLARINET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Lieven Dupont, Principal investigator, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S66825
Record Dates: First submitted 2025-10-23; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Asthma (Diagnosis)
Keywords: Cold air hyperventilation; Asthma diagnosis
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Intervention Model Description: Healthy volunteers will be compared to patients with astma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Healthy volunteers with negative histamine provocation challenge (Other): Healthy volunteers with negative histamine provocation challenge will perform the same tests as the other 2 arms. The healthy volunteers are assigned in this group after the histamine provocation challenge. All will perform one hyperventilation challenge at room temperature (EVH) and one with cold air (CACh) with pre- and post-exposure evaluation on FEV1, respiratory symptoms and local and systemic inflammation
  Interventions: Device: Cold air challenge
- Healthy volunteers with positive histamine provocation challenge (Other): Healthy volunteers with positive histamine provocation challenge will perform the same tests as the other 2 arms. The healthy volunteers are assigned in this group after the histamine provocation challenge. All will perform one hyperventilation challenge at room temperature (EVH) and one with cold air (CACh) with pre- and post-exposure evaluation on FEV1, respiratory symptoms and local and systemic inflammation
  Interventions: Device: Cold air challenge
- Patients with asthma (Other): Patients with asthma will perform the same tests as the other 2 arms. The healthy volunteers are assigned in this group after the histamine provocation challenge. All will perform one hyperventilation challenge at room temperature (EVH) and one with cold air (CACh) with pre- and post-exposure evaluation on FEV1, respiratory symptoms and local and systemic inflammation
  Interventions: Device: Cold air challenge

INTERVENTIONS:
Device: Cold air challenge — This intervention consists of a standardized cold air eucapnic hyperventilation test using a device that controls temperature, humidity, and ventilation. Airway responses are measured via spirometry and biospecimens (serum and sputum supernatant). It is distinguished from other studies by its prospective design and inclusion of both healthy and asthmatic participants
  Other Names: Cold air hyperventilation test

SUMMARY:
In this study, we want to evaluate the feasibility and safety of a CAEH test in healthy volunteers and patients with asthma. We want to develop a CAEH test to differentiate patients with different types of asthma and exercise-induced bronchoconstriction from healthy volunteers and to evaluate whether the respiratory phenotype induced by cold air inhalation differs between subjects with asthma and healthy subjects. Furthermore, we want to evaluate whether the CAEH test is more robust over time compared to the EVH test. Previously, our lab has demonstrated that submaximal exercise at subfreezing temperatures in a climate chamber (-5°C) induces an acute respiratory response in patients with asthma and in healthy subjects who have been exposed to high PM10 (unpublished data). Finally, This study will serve as a preliminary study for a subsequent prospective study in which the results and optimized protocol obtained in this study will be used to further evaluate the feasibility of using this CAEH as a diagnostic tool in asthma compared to EIB (CLARINET2). The present study is required to develop a standardized CAEH test in a safe and feasible manner. This study will also help to identify appropriate endpoints (FEV1, multiple breath washout test, biomarkers…) of the subsequent studies.

DETAILED DESCRIPTION:
In this study, we aim to develop a safe and feasible cold air (-15°C) eucapnic hyperventilation (CAEH) test protocol in which we can compare the lower airway responses between healthy volunteers and subjects with asthma. Consequently, we want to evaluate the effect of cold air inhalation on FEV1, respiratory symptoms, airway integrity, and local and systemic inflammation.

Primary endpoints

The primary endpoint of this study is to compare proportional change in FEV1, (% decrease) after a CAEH test in healthy volunteers and patients with mild to moderate asthma. Post-exposure will be calculated as a time-weighted average over the 30 min after the CAEH test. At each time point (pre-, 5, 10, 15, and 30 minutes post-exposure), FEV1 will be measured in triplicate.

Secondary endpoints

We want to evaluate whether and to what extent the inhalation of cold air during this CAEH test can induce changes in respiratory symptoms (including dyspnea, cough, mucus production, etc.), affects lower airway integrity (airway obstruction (FEV1/FVC), small airway dysfunction (FEF 25/75, lung ventilation inhomogeneity (LCI), bronchial hyperreactivity (PC20 AMP)) and whether it induces (local or systemic) inflammation (different biomarkers in sputum and blood, as defined in section 5.2).

These changes will be compared between healthy volunteers and predisposed subjects with mild to moderate asthma. The abovementioned responses and the proportional change in FEV1 after the CAEH test will be compared to a standard (21°C room air) eucapnic hyperventilation (EVH) test. Furthermore, we will compare the results obtained in this study to the results obtained in the ALASCAIR study of dr. Tatjana Decaesteker. Finally, the effects of the CAEH will be correlated to the amount of air pollution the subject was exposed to, in the days prior to the test (as this may have an effect on the responses to cold air inhalation in healthy volunteers, as found in the Alascair study (unpublished data)), by means of different questionnaires evaluating life style and exposure to air pollution (SF-36, AQLQ, ACQ, SQUASH,…).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old at time of signing informed consent
* BMI between 18 and 28 kg/cm2
* Ability to give informed consent and to comply with study protocol, in the investigator's judgement
* Non-smoking or ex-smokers for at least 12 months with less than 10 pack years
* Normal spirometry

Group specific:

Histamine positive healthy controls: histamine bronchial challenge test (< 8 mg/ml) at screening Healthy controls: histamine bronchial challenge test (≥ 8 mg/ml) at screening

Patients with asthma:

* Physician-diagnosed asthma for at least 6 months
* Post-bronchodilator FEV1 of ≥ 80% at screening
* Documented airway reversibility either by means of post-bronchodilator reversibility of ≥ 12.% and ≥ 200 ml or in the previous 6 months or by means of documented airway hyperresponsiveness (histamine PC20 < 4 mg/ml) at screening
* Asthma control questionnaire (ACQ) ≤ 1.5
* Regular treatment with ICS with or without LABA (unchanged dose for at least 30 days) at a low or medium dose of ICS

Exclusion Criteria:

* Previous history of intubation or admission to ICU due to asthma
* Severe asthma exacerbation within one month prior to screening visit
* Treatment with oral or systemic steroids within one month prior to screening visit
* Previous treatment with biologics for asthma
* Other major concurrent pulmonary (such as COPD, cystic fibrosis, sarcoidosis, interstitial lung disease, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis, bronchiectasis) or cardiovascular disease
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Proportional change in FEV1 after hyperventilation challenge | After each hyperventilation challenge: pre, immediately, 3, 5, 10, 15 and 30 minutes after the challenge
  The proportional change in FEV1 after hyperventilation challenges compared to baseline were measured.

SECONDARY OUTCOMES:
Changes in symptoms | From the first hyperventilation challenge until 1 day after the second
  We want to evaluate changes in respiratory symptoms after challenge. The degree of dyspnea and cough will be determined using BORG scale. This is a 0 to 10 scale.
Lung function changes | After each hyperventilation challenge
  Changes in lung function (FEV1/FVC, FEF25-75, LCI, PEF...) were measured after hyperventilation challenge
Inflammatory parameters | At baseline and after each hyperventilation challenge
  Inflammation was assessed in sputum and blood. Cytokines, allergic response, cellular response, DAMPs and measures of epithelial integrity were assessed.
  Differential cell count will be performed on sputum samples, determining eosinophilic (> 3% eosinophils), neutrophilic (> 61% neutrophils), pauci-granulocytic (< 3% eosinophilic, < 61% neutrophils) and mixed granulocytic (> 3% eosinophilic, > 61% neutrophils). Cytokines will be determined in sputum supernatant with a U-plex assay. Airway inflammation is determined with FeNO. < 25 ppm = eosinophilic inflammation less likely, between 25 - 50 ppm = need further interpretation with additional information and > 50 ppm = indication of eosinophilic airway inflammation. Systemic inflammation will be measured in serum using U-plex assay. allergic response is measured with skin prick automated test on 10 allergens and in serum with total IgE.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Dupont, Principal Investigator — KU Leuven/UZ Leuven
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No